CLINICAL TRIAL: NCT05761925
Title: The COMA Family Program: A Skills-Based Resiliency Program for Caregivers of Patients With Severe Acute Brain Injuries (COMA-F)
Brief Title: The COMA Family Program: A Skills-Based Resiliency Program for Caregivers of Patients With Severe Acute Brain Injuries
Acronym: COMA-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Associate Professor/Director, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021P000423
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Coma; Emotional Distress
Keywords: Severe Acute Brain Injury; Emotional Distress
MeSH Terms: conditions — Coma; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Caregivers will participate in 6 30-minute skills sessions. A clinical psychologist will deliver all of the sessions. The main intervention goal is to provide dyads with resiliency skills to reduce emotional distress and prevent chronic distress.
  Interventions: Behavioral: COMA-F

INTERVENTIONS:
Behavioral: COMA-F — The intervention will teach resiliency skills (mindfulness, coping, interpersonal communication, etc.) to the comatose patient's caregiver. These sessions will take place in person or on Zoom, depending on the participant's preference.

SUMMARY:
The purpose of this study is to pilot a psychosocial skills-based intervention for caregivers of patients with severe acute brain injuries. The data the investigators gather in this study will be used to further refine our COMA-F intervention.

DETAILED DESCRIPTION:
The goal of this study is to refine our proposed intervention (COMA-F) through an open pilot. The investigators will deliver an open pilot of the intervention (N=15 caregivers) to evaluate initial feasibility and acceptability using exit interviews and pre-post assessments.

The open pilot will take place at the Massachusetts General Hospital, University of North Carolina School of Medicine, and University of Maryland School of Medicine neurological intensive care units (NICUs) or step-down units using our established methodology successfully implemented during our previous R21 of our Recovering Together study. Study clinicians will deliver 6, 30 minute sessions of the intervention (at bedside or on Zoom, depending on participant preference). All participants will complete measures at baseline, and after completion of program (6 weeks). They will also complete measures of emotional distress weekly. At the completion of the program, participants will engage in a 5-10 minute exit interview where they will provide feedback of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Eligible caregivers must be caregivers of patients considered to have severe acute brain injury and be unable to communicate with their loved one or clinical team due to their incapacitated nature. Caregivers must meet the following inclusion criteria:

1. Age 18 or older
2. English-speaking
3. Confirmed by the primary clinical team as the primary caregiver for a patient who:

   a. Is age 18 or older; b. Has been admitted to the ICU with a severe acute brain injury: i. Ischemic stroke ii. Intracerebral hemorrhage iii. Subarachnoid hemorrhage iv. Traumatic brain injury v. Hypoxic-ischemic encephalopathy; c. In the judgment of the medical team, has had a Glasgow Coma Scale score below 9 while not intubated OR an inability to following meaningful commands while intubated at any point during his or her hospitalization course for greater than 24 consecutive hours, felt to be due to the brain injury itself and not a confounding factor (i.e., sedation, seizures, etc.); d. Is still alive in the ICU at the time that the clinical team approaches the primary caregiver about possible recruitment; e. Has a prognosis for survival of greater than 3 months and does not have a concurrent diagnosis of a terminal illness or injury, as judged by the clinical team.

   Exclusion Criteria:

   Patient has terminal diagnosis

   Caregiver has:
   * Lack of access to internet and/or a device with a camera
   * Current untreated or unstable severe mental health conditions like bipolar disorder, schizophrenia, or active substance use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Preliminary feasibility of recruitment | 0 weeks
  We will assess the proportion of caregivers enrolled from the number of caregivers eligible.
Preliminary feasibility of assessments | Change from pre-test (0 weeks) to post-test (6 weeks).
  We will assess the proportion of caregivers enrolled that completed all assessments.
Preliminary feasibility of adherence | Change from pre-test (0 weeks) to post-test (6 weeks).
  We will assess the proportion of enrolled caregivers that complete 4 out of 6 sessions.
Preliminary feasibility of therapist fidelity | Change from pre-test (0 weeks) to post-test (6 weeks).
  We will assess the number of sessions in which the therapist adhered 100% to the treatment manual based on a fidelity checklist.
Preliminary treatment satisfaction | post-test (6 weeks after session 1)
  We will assess the proportion of enrolled caregivers that score above the midpoint on the Client Satisfaction Questionnaire-3. Scores range from 3 to 12; higher values indicate greater satisfaction.
Preliminary treatment credibility | post-test (6 weeks after session 1)
  We will use the Credibility and Expectancy Questionnaire (CEQ) to assesses caregivers perceptions that the treatment will work after learning about the study. Scores range from 3-27; higher ratings indicate more belief that the program is logical and will help with the intended outcome.

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Change from pre-test (0 weeks) to post-test (6 weeks)
  We will use the Hospital Anxiety and Depression Scale HADS, a 14-item measure that assesses symptoms of emotional distress (anxiety and depression). The anxiety and depression sub-scale are each scored from 0-21, with higher scores indicating greater severity of symptoms. Scores can be summed to create a global emotional distress score (0-42).
Posttraumatic Stress Disorder Checklist-5 | Change from pre-test (0 weeks) to post-test (6 weeks)
  Post-Traumatic Stress Disorder Checklist - 5; range 0-80, higher scores indicate greater posttraumatic stress
Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | Change from pre-test (0 weeks) to post-test (6 weeks)
  Cognitive and Affective Mindfulness Scale-R (CAMS-R); 12-48, higher scores indicate greater perceived mindfulness
Measure of Current Status Part A (MOCS-A) | Change from pre-test (0 weeks) to post-test (6 weeks)
  Measure of Current Status Part A (MOCS-A); 0-52; higher scores indicate greater perceived ability to cope
Toronto Mindfulness Scale-Trait (TMS-Trait) | Change from pre-test (0 weeks) to post-test (6 weeks)
  Toronto Mindfulness Scale-Trait (TMS-Trait); 0-52, higher scores indicate greater perceived mindfulness (specifically curiosity and de-centering)
Enhancing Recovery in Coronary Heart Disease Social Support Instrument (ESSI) | Change from pre-test (0 weeks) to post-test (6 weeks)
  Enhancing Recovery in Coronary Heart Disease Social Support Instrument (ESSI); the ESSI measures the participant's range of social support in their life. Higher scores indicated higher levels of social support. Total scores range from 8 to 34.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hopsital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Presciutti AM, Rochon E, Alvarez-Frank N, Daily J, Silverman E, Motta M, Vranceanu AM, Hwang DY. Multisite Open Pilot Trial of a Resilience Intervention for Caregivers of Patients with Severe Acute Brain Injury: The Coma Family Program. Neurocrit Care. 2025 Sep 25. doi: 10.1007/s12028-025-02387-x. Online ahead of print. PMID 40999289
- [Derived] Presciutti AM, Woodworth E, Rochon E, Neale M, Motta M, Piazza J, Vranceanu AM, Hwang DY. A Mindfulness-Based Resiliency Program for Caregivers of Patients With Severe Acute Brain Injury Transitioning Out of Critical Care: Protocol for an Open Pilot Trial. JMIR Res Protoc. 2023 Oct 25;12:e50860. doi: 10.2196/50860. PMID 37878376